CLINICAL TRIAL: NCT03327064
Title: A Biomarker Evaluation Trial of UAB30 in Renal Transplant Recipients at High Risk for Non-melanoma Skin Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: COVID-19 pandemic, unable to enroll participants
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Craig Elmets, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UAB30
Record Dates: First submitted 2017-10-26; First posted 2017-10-31 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Non-melanoma Skin Cancer

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Renal Transplant subjects receiving UAB30 (Active Comparator): Generally healthy renal transplant subjects receive UAB30 for 28 days with increased risk of non-melanoma skin cancer as evidenced by a history of prior squamous or basal cell skin cancer, ongoing or history of actinic keratoses and presence at baseline of at least 8 actinic keratosis on the face, neck, scalp and arms.
  Interventions: Drug: UAB30
- Renal Transplant subjects receiving placebo (Placebo Comparator): Generally healthy renal transplant subjects receive placebo for 28 days with increased risk of non-melanoma skin cancer as evidenced by a history of prior squamous or basal cell skin cancer, ongoing or history of actinic keratoses and presence at baseline of at least 8 actinic keratosis on the face, neck, scalp and arms.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: UAB30 — 9cUAB30 promotes homodimer and heterodimer formation with retinoic acid receptors (RARs), and was shown to inhibit breast tumor development in the N-methyl-N-nitrosourea (MNU)-induced rat mammary gland carcinoma model. The compound has also shown efficacy in rodent models of skin cancer. Dose administration will be 160mg daily for 28 days.
  Arms: Renal Transplant subjects receiving UAB30
Drug: Placebo — This matches the UAB30 in appearance. Frequency of dosing will be daily for 28 days.
  Arms: Renal Transplant subjects receiving placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled biomarker study in renal transplant recipients with actinic damage and a history of basal cell carcinomas and/or cutaneous squamous cell carcinomas. There will be two arms to the study: 1) daily oral UAB30 for 28 days; and 2) daily oral placebo for 28 days. The total duration of the study is anticipated to be 5 years. The hypothesis being tested is that a significantly greater percentage of subjects randomized to oral UAB30 over a period of 28 days will achieve ≥30% reduction in biomarkers of proliferation and ≥30% increase in apoptosis biomarkers than those who receive placebo. Cyclin D1 will serve as the primary biomarker.

This investigation will determine whether subjects randomized to UAB30 have an increase in all trans-retinoic acid responsive genes in the skin compared to those receiving placebo. This will include an examination of target effects of UAB30 by evaluating its effects in vivo in humans on the DNA damage response and Src signaling pathways.

DETAILED DESCRIPTION:
Non-melanoma skin cancers (NMSCs), which include basal cell carcinomas (BCCs) and cutaneous squamous carcinomas (SCCs), are the most common malignancy in the U.S.; it is estimated that >3.5 million new NMSCs this year. This represents a tremendous economic impact on the U.S. healthcare system. Most NMSC are caused by overexposure to ultraviolet radiation, and current methods for their prevention consist of recommendations for limitations to sun exposure and avoidance of indoor tanning beds, the regular application of sunscreens, and a variety of other photoprotective activities. Despite these measures, the incidence of NMSCs continues to rise.

NMSCs are a particular problem for organ transplant recipients (OTRs), who must take medicines to protect against rejection of their transplanted organ. These drugs suppress the host immune response that serves to identify and eliminate mutant and neoplastic keratinocytes before they can progress to clinically apparent cancers. Recent research indicates that these drugs also augment signal transduction pathways involved in skin tumor development. NMSCs develop much more frequently in long-term recipients of renal allografts and once present, they behave more aggressively. In immunosuppressed patients, the risk of developing SCCs is 65250-fold higher than in the general population, and the risk of BCCs is 10-fold greater. The rate of SCC metastases in organ transplant recipients is 7%, which is much higher than the general population. For this reason, there has been great interest in identifying novel agents for chemoprevention, which are suitable for use by OTRs.

There will be two groups to the study. Individuals, aged 18 years or older, who have had a renal transplant but are in otherwise general good health, will be given UAB30 (160 mg/day) and will be compared to individuals, aged 18 years or older, who have had a renal transplant and are in otherwise general good health who are given placebo. All participants must be at increased risk of non-melanoma skin cancer as evidenced by a history of prior squamous or basal cell skin cancer, ongoing or history of actinic keratoses, and the presence, at baseline, of at least eight actinic keratoses on the face, neck, scalp and arms. Subjects will be randomized to 28 days of:

1. UAB30 at 160 mg/day, renal transplant recipients
2. placebo renal transplant recipients

At baseline screening, informed consent will be obtained and skin will be examined for potential non-melanoma skin cancers. Any lesions that are clinically suspicious for non-melanoma skin cancer will be removed per standard of care prior to administration of drug. Actinic keratoses will not be removed during the 28 day study period. Two weeks later, once any lesions clinically suspicious for non-melanoma skin cancer have been removed, renal transplant recipients will be randomized to one of the treatment arms described above. Participants will return at 28 days and 112 days for assessment.

1. At randomization and 28 days, 6mm punch biopsies, or the equivalent deep shave biopsies, will be taken for individual biomarkers from non-sun exposed skin, chronically sun exposed skin, and a pre-identified AK. The chronically sun-exposed skin to be biopsied will be no less than 1 cm from the AK to be biopsied.
2. At baseline, at 28 days and at the end of study AK lesions will be assessed and counted, employing techniques that have been validated in other studies.
3. All lesions suspicious for skin cancer will be biopsied and treated appropriately (per standard of care) throughout the study.
4. Adverse events will be assessed, including NMSC and melanoma, from signing of the informed consent through the end of the trial.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age.
* Potential subjects will have at least 8 actinic keratoses (as determined by study dermatologists or qualified designee ).
* ECOG performance status of 0 or 1.
* Participants must have normal organ and marrow function as defined below:
* WBC ≥ 3000/mm3; platelets ≥ 100,000mm3, hemoglobin >10 g/dL
* Bilirubin ≤ upper limit of institutional normal
* Creatinine within institutional normal limits
* Sodium, Potassium, Chloride, Bicarbonate: all ≤ upper limit of institutional normal
* Fasting Triglycerides ≤1.5xULN and Fasting Cholesterol ≤1.5x ULN
* Women of child-bearing potential and men must agree to use two effective forms of birth control prior to study entry and for the duration of study participation and for one month after study completion. Low dose progesterone only birth control pills are not an acceptable form of birth control due to lowered birth control efficacy with retinoids. Males who have had a vasectomy are not considered able to father a child, and therefore are eligible to participate without the use of concurrent birth control. Women who have had a bilateral oophorectomy, hysterectomy, or are greater than 1 year since their last menses, are not considered to be of child-bearing potential, and therefore are eligible to participate without the use of concurrent birth control.

Each of the following is considered to be a single effective method of birth control:

* Combined oral contraceptive pill if used for >30 days prior to entry into the study and continued for 30 days after the last dose of the study agent.
* Implanted hormone if in place for >30 days prior to entry into the study and continued for 30 days after the last dose of the study agent.
* Any implanted device
* Vasectomy
* Tubal ligation
* 2 barrier methods used together
* cervical cap + spermacide or foam
* diaphragm + spermacide or foam
* condom + spermacide or foam
* Females of child-bearing potential must have two negative urine pregnancy tests before starting drug; the first at the time of screening and a second pregnancy test within the first 5 days of their menstrual period.
* Participants must have the ability to understand, and the willingness to sign, a written informed consent document.

Exclusion Criteria:

* Participants may not be taking medications which might interact with UAB30.
* Participants may not be taking lipid lowering agents.
* Participants may not be receiving any other investigational agents.
* Participants with a history of allergic reactions attributed to compounds of similar chemical or biologic composition of retinoids.
* Participants with an uncontrolled intercurrent illness including, but not limited to, ongoing, recurrent or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements. Depression is not exclusionary, but the investigator should make the determination if patients with depression are eligible.
* Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with UAB30, breastfeeding must be discontinued for the duration of study participation and for one month after the last dose of the study agent if the mother is treated with UAB30.
* Individuals known to be HIV-positive may not participate in this study. The uncertain immune status of HIV-positive people and the potential risks of taking part in this study are too great to justify a study with low likelihood of benefit
* Individuals with a history of cancer diagnosis or reoccurrence <5 years from study entry may not participate. However, individuals with a history of squamous or basal cell carcinoma of the skin <5 years from study entry will not be excluded from this study.
* Because of the uncertain risk of UAB30 to unborn fetuses and children, pregnant women and children will not be allowed in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Percent of subjects that achieve at least a 30% reduction in cyclin D1 expression in normal skin, in sun-exposed skin, and in actinic keratoses from baseline to the end of UAB30 administration (day 28) | Baseline to day 28
  Skin biopsies will be performed on normal skin, sun-exposed skin and one actinic keratosis at study initiation and again at day 28. The skin specimens will be processed for immunohistochemistry (IHC), which will be used for cyclin D1 expression. Quantification of cyclin D1 will be performed on microscopic sections by digital image analysis. Cyclin D1 will be measured at randomization (baseline) and after 28 days on UAB30.

SECONDARY OUTCOMES:
Percent of subjects with 30% or greater decrease in proliferation as detected by Ki67 staining | Baseline to day 28
  Skin biopsies will be performed on normal skin, sun-exposed skin and one actinic keratosis at study initiation and again at day 28. The skin specimens will be processed for immunohistochemistry (IHC), which will be used for Ki67 expression. Quantification of Ki67will be performed on microscopic sections by digital image analysis. Ki67 will be measured at randomization and after 28 days on UAB30.
Percent of subjects with 30% or greater decreased proliferation as detected by PCNA staining | Baseline (randomization) to day 28
  Skin biopsies will be performed on normal skin, sun-exposed skin and one actinic keratosis at study initiation and again at day 28. The skin specimens will be processed for immunohistochemistry (IHC), which will be used for PCNA expression as a marker for cellular proliferation. Quantification of PCNA will be performed on microscopic sections by digital image analysis. PCNA will be measured at randomization and after 28 days on UAB30.
Percent of subjects with 30% or greater increased apoptosis as detected by the TUNEL assay | Baseline (randomization) to day 28
  Skin biopsies will be performed on normal skin, sun-exposed skin and one actinic keratosis at study initiation and again at day 28. The skin specimens will be processed for TUNEL assay done by using an in situ cell death detection, fluorescein kit. Quantification of TUNEL positive cells will be performed on microscopic sections by digital image analysis. TUNEL positive cells will be measured at randomization and after 28 days on UAB30.
• Percent of subjects with 30% or greater decreased expression of the apoptotic protein Bcl-2 | Baseline (randomization) to day 28
  Skin biopsies will be performed on normal skin, sun-exposed skin and one actinic keratosis. Protein will be isolated from skin biopsies and the biomarker will be assessed by Western blot analysis. Bcl-2 expression will be measured at randomization and after 28 days on UAB30.
Percent of subjects with 30% or greater increased apoptosis as detected by cleaved caspase 3 | Baseline (randomization) to day 28
  Skin biopsies will be performed on normal skin, sun-exposed skin and one actinic keratosis. Protein will be isolated from skin biopsies and the biomarker will be assessed by Western blot analysis. Cleaved caspase 3 expression will be measured at randomization and after 28 days on UAB30.
Percent of subjects with 30% or greater increase in DNA damage repair as detected by a reduction in γH2AX staining | Baseline (randomization)to day 28
  Skin biopsies will be performed on normal skin, sun-exposed skin and one actinic keratosis. Immunofluorescence will be used to assess γH2AX expression. Quantification of γH2AX positive cells will be performed on microscopic sections by digital image analysis at randomization and after 28 days on UAB30.
Percent of subjects with 30% or greater increased apoptosis as detected by DNA damage repair pathway proteins : p-γH2AX | Baseline (randomization)to day 28
  Skin biopsies will be performed on normal skin, sun-exposed skin and one actinic keratosis. RNA will be isolated from skin biopsies and the biomarkers will be assessed by qPCR. RNA for these biomarkers will be measured at randomization and after 28 days on UAB30
Percent of subjects with 30% or greater increased expression of the phosphorylated form of the DNA repair protein ATM | Baseline (randomization) to day 28
  Skin biopsies will be performed on normal skin, sun-exposed skin and one actinic keratosis. Protein will be isolated from skin biopsies and the biomarker will be assessed by Western blot analysis. Phosphorylated ATM will be measured at randomization and after 28 days on UAB30.
Percent of subjects with 30% or greater enhancement in the phosphorylation of DNA damage response protein ATM. | Baseline (randomization) to day 28
  Skin biopsies will be performed on normal skin, sun-exposed skin and one actinic keratosis. Proteins will be isolated from skin biopsies and the biomarkers will be assessed by Western blot analysis. The phosphorylated proteins will be measured at randomization and after 28 days on UAB30.
Percent of subjects with 30% or greater enhancement in the phosphorylation of DNA damage response protein RAD51. | Baseline (randomization) to day 28
  Skin biopsies will be performed on normal skin, sun-exposed skin and one actinic keratosis. Proteins will be isolated from skin biopsies and the biomarkers will be assessed by Western blot analysis. The phosphorylated proteins will be measured at randomization and after 28 days on UAB30.
Percent of subjects with 30% or greater enhancement in the phosphorylation of DNA damage response protein ATR. | Baseline (randomization) to day 28
  Skin biopsies will be performed on normal skin, sun-exposed skin and one actinic keratosis. Proteins will be isolated from skin biopsies and the biomarkers will be assessed by Western blot analysis. The phosphorylated proteins will be measured at randomization and after 28 days on UAB30.
Percent of subjects with 30% or greater enhancement in the phosphorylation of DNA damage response protein CHK1/2. | Baseline (randomization) to day 28
  Skin biopsies will be performed on normal skin, sun-exposed skin and one actinic keratosis. Proteins will be isolated from skin biopsies and the biomarkers will be assessed by Western blot analysis. The phosphorylated proteins will be measured at randomization and after 28 days on UAB30.
Percent of subjects with 30% or greater enhancement in the phosphorylation of DNA damage response proteins ATR. | Baseline (randomization) to day 28
  Skin biopsies will be performed on normal skin, sun-exposed skin and one actinic keratosis. Proteins will be isolated from skin biopsies and the biomarkers will be assessed by Western blot analysis. The phosphorylated proteins will be measured at randomization and after 28 days on UAB30.
Percent of subjects with 30% or greater decreased numbers of CD4+ T-cellscount | Baseline (randomization) to day 28
  Skin biopsies will be performed on normal skin, sun-exposed skin and one actinic keratosis. The skin specimens will be processed for immunofluorescence, which will be used for CD4+ expression as a marker for immunological parameters. Quantification of CD4+ expression will be performed on microscopic sections by digital image analysis. CD4+ expression will be measured at randomization and after 28 days on UAB30
Percent of subjects with 30% or greater increased numbers of CD8+ T-cells | Baseline (randomization) to day 28
  Skin biopsies will be performed on normal skin, sun-exposed skin and one actinic keratosis. The skin specimens will be processed for immunofluorescence, which will be used for CD8+ expression as a marker for immunological parameters. Quantification of CD8+ expression will be performed on microscopic sections by digital image analysis. CD8+ expression will be measured at randomization and after 28 days on UAB30
Percent of subjects with 30% or greater change in all trans-retinoic acid target genes : (ATRA) responsive genes (DHRS3, STRA6, MUC21, GABRP, DHRS9) | Baseline (randomization) to day 28
  Skin biopsies will be performed on normal skin, sun-exposed skin and one actinic keratosis. RNA will be isolated from skin biopsies and the biomarker will be assessed by qPCR. RNA for these biomarkers will be measured at randomization and after 28 days on UAB30
Percent of subjects with 30% or greater decreased expression of the immunological marker for regulatory T-cells, FoxP3 | Baseline (randomization) to day 28
  Skin biopsies will be performed on normal skin, sun-exposed skin and one actinic keratosis. RNA will be isolated from skin biopsies and the biomarker will be assessed by qPCR. RNA for this biomarkers will be measured at randomization and after 28 days on UAB30
Percent of subjects with 30% or greater increased expression of the immunological marker for regulatory T-cells: IFN-γ | Baseline (randomization) to day 28
  Skin biopsies will be performed on normal skin, sun-exposed skin and one actinic keratosis. RNA will be isolated from skin biopsies and the biomarkers will be assessed by qPCR. RNA for these biomarkers will be measured at randomization and after 28 days on UAB30
Percent of subjects with 30% or greater increased expression of the immunological marker for regulatory T-cells: IL-10 | Baseline (randomization) to day 28
  Skin biopsies will be performed on normal skin, sun-exposed skin and one actinic keratosis. RNA will be isolated from skin biopsies and the biomarker will be assessed by qPCR. RNA for these biomarkers will be measured at randomization and after 28 days on UAB30
Percent of subjects with 30% or greater increased expression of the immunological marker for Th17 cells. | Baseline (randomization) to day 28
  Skin biopsies will be performed on normal skin, sun-exposed skin and one actinic keratosis. RNA will be isolated from skin biopsies and the biomarkers will be assessed by qPCR. RNA for these biomarkers will be measured at randomization and after 28 days on UAB30.
Percent of subjects with 30% or greater decreased proliferation as detected by genes associated with immunological parameters: IL-22 | Baseline (randomization) to day 28
  Skin biopsies will be performed on normal skin, sun-exposed skin and one actinic keratosis. RNA will be isolated from skin biopsies and the biomarkers will be assessed by qPCR. RNA for these biomarkers will be measured at randomization and after 28 days on UAB30
Number of subjects in each group with actinic keratosis at the end of treatment with UAB30 (day 28) and 84 days after the end of treatment with UAB30 (day 112). | Baseline (randomization) to day 112
  AKs will be counted and recorded at randomization, after 28 days on UAB30 and 84 days later (day 112). At the end of the study, new, persistent and regressed AKs will be recorded. Total number of AKs, number of new AKs, and number of regressed AKs will be assessed.
Mean number of toxicities experienced by subjects in each group treatment with UAB30 without signs of significant toxicity in organ transplant recipients.. | baseline to day 28
  For all subjects the mean number of toxicities (grade 3 or 4) per subject will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Craig Elmets, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Dermatology, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No